CLINICAL TRIAL: NCT00005146
Title: Diabetes and Cardiovascular Risk In Mexico City (San Antonio Heart Study)
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1017; R01HL024799 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Diabetes Mellitus, Non-insulin Dependent; Diabetes Mellitus
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine factors beyond obesity which contribute to diabetes and cardiovascular risk in Mexicans and Mexican Americans. To test the hypothesis that at any given level of adiposity Mexican Americans will be more insulin resistant than Anglos and that the insulin resistance in Mexican Americans is proportional to the degree of Native American ancestry.

DETAILED DESCRIPTION:
BACKGROUND:

The present study was preceded by the earlier San Antonio Heart Study 1 supported under this grant. The San Antonio Heart Study 1 was a population-based survey of diabetes and cardiovascular risk factors in Mexican American and non-Hispanic whites conducted from 1979 to 1982. Participants included all men and non-pregnant women ages 24 to 64, who resided in households randomly sampled from three socio-culturally distinct neighborhoods of San Antonio. The low-income barrio residents were almost exclusively traditional Mexican-Americans. The middle-income neighborhood was ethnically balanced with equal numbers of Mexican Americans and Anglos whereas the upper income suburb was approximately 90 percent Anglo. Risk factors measured included obesity, glucose intolerance, hypertriglyceridemia, low levels of high density lipoprotein cholesterol, and blood pressure. The total number of people who were examined medically was 2,386, divided as follows: 1,288 Mexican Americans; 929 Anglos; and 169 other Hispanics such as Cubans. The San Antonio Heart Study was designed to test the hypothesis that as Mexican Americans became progressively more affluent and acculturated to 'mainstream' United States culture, they would gradually lose their diabetic pattern of cardiovascular risk factors of obesity, diabetes, and hypertriglyceridemia.

DESIGN NARRATIVE:

Beginning in 1979, a random sample was conducted to select participants. Sampling was performed to match the two groups on obesity, thereby enabling an analysis of the ethnic differences in diabetes and cardiovascular risk factors independent of the confounding effects of obesity. For those selected, an interview and medical examination were conducted in a mobile clinic. The interview consisted of a personal and family history of diabetes and cardiovascular risk, knowledge of and attitudes towards cardiovascular risk factors, dietary questionnaire, Rose Angina questionnaire, intermittent claudication questionnaire, and medication history. The medical examination consisted of anthropometric measurements, plasma glucose, plasma insulin, hemoglobin, serum cholesterol, triglyceride, HDL, LDL, and VLDL, genetic markers, blood pressure, skin color and electrocardiogram. It was estimated that 400 diabetics would be available over the four years of the study to permit a Diabetic Recall Examination. The purpose of the Diabetic Recall Examination was to assess possible end-organ complications of diabetes involving the eye, kidney, peripheral and autonomic nervous systems, and the peripheral vascular system. The assessment provided baseline data on diabetics which was used for a prospective incidence study. Beginning in 1989, a prevalence survey of type II diabetes mellitus and cardiovascular risk factors was conducted in a low-income barrio in Mexico City. Information collected on this population included demographic data, socioeconomic status, level of acculturation, medical history, diet, exercise, and smoking. The physical examination included measurements of blood pressure, obesity, body fat distribution, and skin color. The laboratory examination included measurements of lipids and lipoproteins, oral glucose tolerance tests, fasting and post-glucose load insulin concentrations and genetic markers.

Beginning in FY 1989, Michael Stern and associates carried out an epidemiologic study of type II diabetes mellitus and cardiovascular risk factors in a low-income barrio of Mexico City and compared results to those obtained in San Antonio. They recruited and interviewed subjects for data on demographics, socioeconomic status, level of acculturation, medical history, health habits including diet, physical exercise, and smoking. The physical examination included blood pressure, obesity, body fat distribution, skin color, the latter to estimate percent Native American genetic admixture. The laboratory examination included measurements of lipids and lipoproteins, an oral glucose tolerance test to determine the prevalence of diabetes according to the National Diabetes Data Group criteria, fasting and post-glucose load insulin concentrations, and genetic markers.

The study was renewed in 1996 through August, 2001. A 3.25 year followup examination (FU1) of a cohort of 2,296 Mexican men and women, ages 35-64 years at baseline, was completed. The cohort was re-examined at 3.25-year intervals (6.5 years (FU2) and 9.75 years (FU3) after baseline). The investigators tested the hypothesis that different risk factors would prevail in the early (more than 3.25 years prior to conversion to diabetes) than in the late (3.25 years or less prior to conversion) prediabetic period. They hypothesized that in the early prediabetic period risk factors associated with the Insulin Resistance Syndrome would predominate, i.e., high "specific" insulin concentration (measured by a specific immunoassay), hypertriglyceridemia, low HDL-cholesterol, and hypertension, whereas in the late prediabetic period factors associated with insulin secretory failure, i.e., increased proinsulin and low "specific" insulin, would predominate.

Michael Stern and associates assessed carotid wall thickness by ultrasonography on all subjects at FU1 and planned to repeat this at FU2. They measured advanced glycation endproduct (AGE)-modified apolipoprotein B and a panel of inflammatory risk factors (serum albumin, serum amyloid A, alpha1-acid glycoprotein, and C-reactive protein) on stored contingency specimens from baseline and FU1 in order to determine if these factors predicted accelerated thickening of carotid walls and/or the development of type II diabetes. They also quantified the extent to which carotid wall thickness and ECG documented myocardial infarction preceded clinical diabetes as predicted by the "common soil" hypothesis, i.e., the hypothesis that both type II diabetes and atherosclerosis have common genetic and environmental antecedents.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1979-05; Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stern — University of Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stern MP, Pugh JA, Gaskill SP, Hazuda HP. Knowledge, attitudes, and behavior related to obesity and dieting in Mexican Americans and Anglos: the San Antonio Heart Study. Am J Epidemiol. 1982 Jun;115(6):917-28. doi: 10.1093/oxfordjournals.aje.a113379. PMID 7091149
- [Background] Stern MP, Gaskill SP, Hazuda HP, Gardner LI, Haffner SM. Does obesity explain excess prevalence of diabetes among Mexican Americans? Results of the San Antonio Heart Study. Diabetologia. 1983 Apr;24(4):272-7. doi: 10.1007/BF00282712. PMID 6862133
- [Background] Malina RM, Little BB, Stern MP, Gaskill SP, Hazuda HP. Ethnic and social class differences in selected anthropometric characteristics of Mexican American and Anglo adults: the San Antonio Heart Study. Hum Biol. 1983 Dec;55(4):867-83. No abstract available. PMID 6674108
- [Background] Relethford JH, Stern MP, Gaskill SP, Hazuda HP. Social class, admixture, and skin color variation in Mexican-Americans and Anglo-Americans living in San Antonio, Texas. Am J Phys Anthropol. 1983 May;61(1):97-102. doi: 10.1002/ajpa.1330610110. PMID 6869517
- [Background] Hazuda HP, Stern MP, Gaskill SP, Haffner SM, Gardner LI. Ethnic differences in health knowledge and behaviors related to the prevention and treatment of coronary heart disease. The San Antonio Heart Study. Am J Epidemiol. 1983 Jun;117(6):717-28. doi: 10.1093/aje/117.6.717. PMID 6859027
- [Background] Haffner SM, Rosenthal M, Hazuda HP, Stern MP, Franco LJ. Evaluation of three potential screening tests for diabetes mellitus in a biethnic population. Diabetes Care. 1984 Jul-Aug;7(4):347-53. doi: 10.2337/diacare.7.4.347. PMID 6468231
- [Background] Gardner LI Jr, Stern MP, Haffner SM, Gaskill SP, Hazuda HP, Relethford JH, Eifler CW. Prevalence of diabetes in Mexican Americans. Relationship to percent of gene pool derived from native American sources. Diabetes. 1984 Jan;33(1):86-92. doi: 10.2337/diab.33.1.86. PMID 6690348
- [Background] Stern MP, Rosenthal M, Haffner SM, Hazuda HP, Franco LJ. Sex difference in the effects of sociocultural status on diabetes and cardiovascular risk factors in Mexican Americans. The San Antonio Heart Study. Am J Epidemiol. 1984 Dec;120(6):834-51. doi: 10.1093/oxfordjournals.aje.a113956. PMID 6507426
- [Background] Deyo RA, Diehl AK, Hazuda H, Stern MP. A simple language-based acculturation scale for Mexican Americans: validation and application to health care research. Am J Public Health. 1985 Jan;75(1):51-5. doi: 10.2105/ajph.75.1.51. PMID 3966599
- [Background] Rosenthal M, McMahan CA, Stern MP, Eifler CW, Haffner SM, Hazuda HP, Franco LJ. Evidence of bimodality of two hour plasma glucose concentrations in Mexican Americans: results from the San Antonio Heart study. J Chronic Dis. 1985;38(1):5-16. doi: 10.1016/0021-9681(85)90003-7. PMID 3972950
- [Background] Haffner SM, Knapp JA, Stern MP, Hazuda HP, Rosenthal M, Franco LJ. Coffee consumption, diet, and lipids. Am J Epidemiol. 1985 Jul;122(1):1-12. doi: 10.1093/oxfordjournals.aje.a114067. PMID 4014187
- [Background] Franco LJ, Stern MP, Rosenthal M, Haffner SM, Hazuda HP, Comeaux PJ. Prevalence, detection, and control of hypertension in a biethnic community. The San Antonio Heart Study. Am J Epidemiol. 1985 May;121(5):684-96. doi: 10.1093/aje/121.5.684. PMID 4014160
- [Background] Knapp JA, Haffner SM, Young EA, Hazuda HP, Gardner L, Stern MP. Dietary intakes of essential nutrients among Mexican-Americans and Anglo-Americans: the San Antonio Heart Study. Am J Clin Nutr. 1985 Aug;42(2):307-16. doi: 10.1093/ajcn/42.2.307. PMID 4025200
- [Background] Stern MP: Diabetes in Hispanic Americans. In: Diabetes in America Harris MI, Hamman R (Eds). U.S. Government Printing Office, NIH Publication No. 85-1468, Washington DC, pp IX-1-11, Aug 1985
- [Background] Stern MP, Rosenthal M, Haffner SM. A new concept of impaired glucose tolerance. Relation to cardiovascular risk. Arteriosclerosis. 1985 Jul-Aug;5(4):311-4. doi: 10.1161/01.atv.5.4.311. No abstract available. PMID 4015505
- [Background] Diehl AK, Rosenthal M, Hazuda HP, Comeaux PJ, Stern MP. Socioeconomic status and the prevalence of clinical gallbladder disease. J Chronic Dis. 1985;38(12):1019-26. doi: 10.1016/0021-9681(85)90100-6. PMID 3877735
- [Background] Haffner SM, Knapp JA, Hazuda HP, Stern MP, Young EA. Dietary intakes of macronutrients among Mexican Americans and Anglo Americans: the San Antonio heart study. Am J Clin Nutr. 1985 Dec;42(6):1266-75. doi: 10.1093/ajcn/42.6.1266. PMID 4072960
- [Background] Hazuda HP, Comeaux PJ, Stern MP, Haffner SM, Eifler CW, Rosenthal M. A comparison of three indicators for identifying Mexican Americans in epidemiologic research. Methodological findings from the San Antonio Heart Study. Am J Epidemiol. 1986 Jan;123(1):96-112. doi: 10.1093/oxfordjournals.aje.a114228. PMID 3940446
- [Background] Haffner SM, Stern MP, Hazuda HP, Rosenthal M, Knapp JA, Malina RM. Role of obesity and fat distribution in non-insulin-dependent diabetes mellitus in Mexican Americans and non-Hispanic whites. Diabetes Care. 1986 Mar-Apr;9(2):153-61. doi: 10.2337/diacare.9.2.153. PMID 3698781
- [Background] Haffner SM, Stern MP, Hazuda HP, Rosenthal M, Knapp JA. The role of behavioral variables and fat patterning in explaining ethnic differences in serum lipids and lipoproteins. Am J Epidemiol. 1986 May;123(5):830-9. doi: 10.1093/oxfordjournals.aje.a114312. PMID 3962965
- [Background] Hazuda HP, Haffner SM, Stern MP, Knapp JA, Eifler CW, Rosenthal M. Employment status and women's protection against coronary heart disease. Findings from the San Antonio Heart Study. Am J Epidemiol. 1986 Apr;123(4):623-40. doi: 10.1093/oxfordjournals.aje.a114282. PMID 3953541
- [Background] Stern MP, Ferrell RE, Rosenthal M, Haffner SM, Hazuda HP. Association between NIDDM, RH blood group, and haptoglobin phenotype. Results from the San Antonio Heart Study. Diabetes. 1986 Apr;35(4):387-91. doi: 10.2337/diab.35.4.387. PMID 3082699
- [Background] Stern MP, Haffner SM. Body fat distribution and hyperinsulinemia as risk factors for diabetes and cardiovascular disease. Arteriosclerosis. 1986 Mar-Apr;6(2):123-30. doi: 10.1161/01.atv.6.2.123. PMID 3513749
- [Background] Haffner SM, Stern MP, Hazuda HP, Pugh JA, Patterson JK. Hyperinsulinemia in a population at high risk for non-insulin-dependent diabetes mellitus. N Engl J Med. 1986 Jul 24;315(4):220-4. doi: 10.1056/NEJM198607243150403. PMID 3523246
- [Background] Haffner SM, Stern MP, Hazuda HP, Pugh J, Patterson JK, Malina R. Upper body and centralized adiposity in Mexican Americans and non-Hispanic whites: relationship to body mass index and other behavioral and demographic variables. Int J Obes. 1986;10(6):493-502. PMID 3804566
- [Background] Chakraborty R, Ferrell RE, Stern MP, Haffner SM, Hazuda HP, Rosenthal M. Relationship of prevalence of non-insulin-dependent diabetes mellitus to Amerindian admixture in the Mexican Americans of San Antonio, Texas. Genet Epidemiol. 1986;3(6):435-54. doi: 10.1002/gepi.1370030608. PMID 3803913
- [Background] Haffner SM, Stern MP, Hazuda HP, Pugh J, Patterson JK. Do upper-body and centralized adiposity measure different aspects of regional body-fat distribution? Relationship to non-insulin-dependent diabetes mellitus, lipids, and lipoproteins. Diabetes. 1987 Jan;36(1):43-51. doi: 10.2337/diab.36.1.43. PMID 3792664
- [Background] Diehl AK, Haffner SM, Hazuda HP, Stern MP. Coronary risk factors and clinical gallbladder disease: an approach to the prevention of gallstones? Am J Public Health. 1987 Jul;77(7):841-5. doi: 10.2105/ajph.77.7.841. PMID 3496013
- [Background] Haffner SM. Hyperinsulinemia as a possible etiology for the high prevalence of non insulin dependent diabetes in Mexican Americans. Diabete Metab. 1987 Jul;13(3 Pt 2):337-44. PMID 3308561
- [Background] Knapp JA, Hazuda HP, Haffner SM, Young EA, Stern MP. A saturated fat/cholesterol avoidance scale: sex and ethnic differences in a biethnic population. J Am Diet Assoc. 1988 Feb;88(2):172-7. PMID 3339203
- [Background] Haffner SM, Fong D, Hazuda HP, Pugh JA, Patterson JK. Hyperinsulinemia, upper body adiposity, and cardiovascular risk factors in non-diabetics. Metabolism. 1988 Apr;37(4):338-45. doi: 10.1016/0026-0495(88)90133-3. PMID 3282148
- [Background] Haffner SM, Fong D, Stern MP, Pugh JA, Hazuda HP, Patterson JK, van Heuven WA, Klein R. Diabetic retinopathy in Mexican Americans and non-Hispanic whites. Diabetes. 1988 Jul;37(7):878-84. doi: 10.2337/diab.37.7.878. PMID 3384186
- [Background] Haffner SM, Katz MS, Stern MP, Dunn JF. The relationship of sex hormones to hyperinsulinemia and hyperglycemia. Metabolism. 1988 Jul;37(7):683-8. doi: 10.1016/0026-0495(88)90091-1. PMID 3290626
- [Background] Haffner SM, Katz MS, Stern MP, Dunn JF. Relationship of sex hormone binding globulin to overall adiposity and body fat distribution in a biethnic population. Int J Obes. 1989;13(1):1-9. PMID 2703288
- [Background] Pugh JA, Stern MP, Haffner SM, Hazuda HP, Patterson J. Detection and treatment of hypercholesterolemia in a biethnic community, 1979-1985. J Gen Intern Med. 1988 Jul-Aug;3(4):331-6. doi: 10.1007/BF02595790. PMID 3404294
- [Background] Stern MP, Haffner SM. Do anthropometric differences between Mexican Americans and non-Hispanic whites explain ethnic differences in metabolic variables? Acta Med Scand Suppl. 1988;723:37-44. doi: 10.1111/j.0954-6820.1987.tb05926.x. No abstract available. PMID 3164973
- [Background] Haffner SM, Stern MP, Hazuda HP, Mitchell BD, Patterson JK. Increased insulin concentrations in nondiabetic offspring of diabetic parents. N Engl J Med. 1988 Nov 17;319(20):1297-301. doi: 10.1056/NEJM198811173192001. PMID 3054549
- [Background] Hazuda HP, Haffner SM, Stern MP, Eifler CW. Effects of acculturation and socioeconomic status on obesity and diabetes in Mexican Americans. The San Antonio Heart Study. Am J Epidemiol. 1988 Dec;128(6):1289-301. doi: 10.1093/oxfordjournals.aje.a115082. PMID 3195568
- [Background] Haffner SM, Katz MS, Stern MP, Dunn JF. Association of decreased sex hormone binding globulin and cardiovascular risk factors. Arteriosclerosis. 1989 Jan-Feb;9(1):136-43. doi: 10.1161/01.atv.9.1.136. PMID 2643424
- [Background] Diehl AK, Stern MP. Special health problems of Mexican-Americans: obesity, gallbladder disease, diabetes mellitus, and cardiovascular disease. Adv Intern Med. 1989;34:73-96. No abstract available. PMID 2644769
- [Background] Haffner SM, Diehl AK, Stern MP, Hazuda HP. Central adiposity and gallbladder disease in Mexican Americans. Am J Epidemiol. 1989 Mar;129(3):587-95. doi: 10.1093/oxfordjournals.aje.a115171. PMID 2916552
- [Background] Haffner SM, Hazuda HP, Stern MP, Patterson JK, Van Heuven WA, Fong D. Effects of socioeconomic status on hyperglycemia and retinopathy levels in Mexican Americans with NIDDM. Diabetes Care. 1989 Feb;12(2):128-34. doi: 10.2337/diacare.12.2.128. PMID 2702895
- [Background] Stern MP, Patterson JK, Haffner SM, Hazuda HP, Mitchell BD. Lack of awareness and treatment of hyperlipidemia in type II diabetes in a community survey. JAMA. 1989 Jul 21;262(3):360-4. PMID 2739037
- [Background] Raboudi SH, Mitchell BD, Stern MP, Eifler CW, Haffner SM, Hazuda HP, Frazier ML. Type II diabetes mellitus and polymorphism of insulin-receptor gene in Mexican Americans. Diabetes. 1989 Aug;38(8):975-80. doi: 10.2337/diab.38.8.975. PMID 2568958
- [Background] Haffner SM, Mitchell BD, Pugh JA, Stern MP, Kozlowski MK, Hazuda HP, Patterson JK, Klein R. Proteinuria in Mexican Americans and non-Hispanic whites with NIDDM. Diabetes Care. 1989 Sep;12(8):530-6. doi: 10.2337/diacare.12.8.530. PMID 2776587
- [Background] Diehl AK, Haffner SM, Knapp JA, Hazuda HP, Stern MP. Dietary intake and the prevalence of gallbladder disease in Mexican Americans. Gastroenterology. 1989 Dec;97(6):1527-33. doi: 10.1016/0016-5085(89)90399-5. PMID 2583417
- [Background] Haffner SM, Stern MP, Hazuda HP, Mitchell BD, Patterson JK, Ferrannini E. Parental history of diabetes is associated with increased cardiovascular risk factors. Arteriosclerosis. 1989 Nov-Dec;9(6):928-33. doi: 10.1161/01.atv.9.6.928. PMID 2686606
- [Background] Haffner SM, Karhapaa P, Rainwater DL, Mykkanen L, Aldrete G Jr, Laakso M. Insulin sensitivity and Lp(a) concentrations in normoglycemic men. Diabetes Care. 1995 Feb;18(2):193-9. doi: 10.2337/diacare.18.2.193. PMID 7729297
- [Background] Haffner SM, Miettinen H, Stern MP. Insulin secretion and resistance in nondiabetic Mexican Americans and non-Hispanic whites with a parental history of diabetes. J Clin Endocrinol Metab. 1996 May;81(5):1846-51. doi: 10.1210/jcem.81.5.8626845.
- [Background] Haffner SM, Stern MP, Mitchell BD, Hazuda HP, Patterson JK. Incidence of type II diabetes in Mexican Americans predicted by fasting insulin and glucose levels, obesity, and body-fat distribution. Diabetes. 1990 Mar;39(3):283-8. doi: 10.2337/diab.39.3.283. PMID 2407581
- [Background] Haffner SM, Mitchell BD, Stern MP, Hazuda HP, Patterson JK. Public health significance of upper body adiposity for non-insulin dependent diabetes mellitus in Mexican Americans. Int J Obes Relat Metab Disord. 1992 Mar;16(3):177-84. PMID 1317826
- [Background] Jameel N, Pugh JA, Mitchell BD, Stern MP. Dietary protein intake is not correlated with clinical proteinuria in NIDDM. Diabetes Care. 1992 Feb;15(2):178-83. doi: 10.2337/diacare.15.2.178. PMID 1547674
- [Background] Haffner SM, Dunn JF, Katz MS. Relationship of sex hormone-binding globulin to lipid, lipoprotein, glucose, and insulin concentrations in postmenopausal women. Metabolism. 1992 Mar;41(3):278-84. doi: 10.1016/0026-0495(92)90271-b. PMID 1542267
- [Background] Haffner SM, Mitchell BD, Stern MP, Hazuda HP. Macrovascular complications in Mexican Americans with type II diabetes. Diabetes Care. 1991 Jul;14(7):665-71. doi: 10.2337/diacare.14.7.665. PMID 1914816
- [Background] Stern MP, Knapp JA, Hazuda HP, Haffner SM, Patterson JK, Mitchell BD. Genetic and environmental determinants of type II diabetes in Mexican Americans. Is there a "descending limb" to the modernization/diabetes relationship? Diabetes Care. 1991 Jul;14(7):649-54. doi: 10.2337/diacare.14.7.649. PMID 1914814
- [Background] Ferrannini E, Haffner SM, Stern MP, Mitchell BD, Natali A, Hazuda HP, Patterson JK. High blood pressure and insulin resistance: influence of ethnic background. Eur J Clin Invest. 1991 Jun;21(3):280-7. doi: 10.1111/j.1365-2362.1991.tb01371.x. PMID 1909631
- [Background] Haffner SM, Katz MS, Dunn JF. Increased upper body and overall adiposity is associated with decreased sex hormone binding globulin in postmenopausal women. Int J Obes. 1991 Jul;15(7):471-8. PMID 1894424
- [Background] Ferrannini E, Haffner SM, Mitchell BD, Stern MP. Hyperinsulinaemia: the key feature of a cardiovascular and metabolic syndrome. Diabetologia. 1991 Jun;34(6):416-22. doi: 10.1007/BF00403180. PMID 1884900
- [Background] Stern MP. Kelly West Lecture. Primary prevention of type II diabetes mellitus. Diabetes Care. 1991 May;14(5):399-410. doi: 10.2337/diacare.14.5.399. PMID 2060452
- [Background] Hazuda HP, Mitchell BD, Haffner SM, Stern MP. Obesity in Mexican American subgroups: findings from the San Antonio Heart Study. Am J Clin Nutr. 1991 Jun;53(6 Suppl):1529S-1534S. doi: 10.1093/ajcn/53.6.1529S. PMID 2031483
- [Background] Haffner SM, Klein R, Dunn JF, Moss SE, Klein BE. Increased testosterone in type I diabetic subjects with severe retinopathy. Ophthalmology. 1990 Oct;97(10):1270-4. doi: 10.1016/s0161-6420(90)32428-4. PMID 2147054
- [Background] Haffner SM, Katz MS, Dunn JF. The relationship of insulin sensitivity and metabolic clearance of insulin to adiposity and sex hormone binding globulin. Endocr Res. 1990;16(3):361-76. doi: 10.1080/07435809009033012. PMID 2292238
- [Background] Berkus MD, Stern MP, Mitchell BD, Newton ER, Langer O. Does fasting interval affect the glucose challenge test? Am J Obstet Gynecol. 1990 Dec;163(6 Pt 1):1812-7. doi: 10.1016/0002-9378(90)90755-v. PMID 2256487
- [Background] Haffner SM, Stern MP, Dunn J, Mobley M, Blackwell J, Bergman RN. Diminished insulin sensitivity and increased insulin response in nonobese, nondiabetic Mexican Americans. Metabolism. 1990 Aug;39(8):842-7. doi: 10.1016/0026-0495(90)90130-5. PMID 2198435
- [Background] Haffner SM, Diehl AK, Mitchell BD, Stern MP, Hazuda HP. Increased prevalence of clinical gallbladder disease in subjects with non-insulin-dependent diabetes mellitus. Am J Epidemiol. 1990 Aug;132(2):327-35. doi: 10.1093/oxfordjournals.aje.a115662. PMID 2196792
- [Background] Haffner SM, Stern MP, Gruber MK, Hazuda HP, Mitchell BD, Patterson JK. Microalbuminuria. Potential marker for increased cardiovascular risk factors in nondiabetic subjects? Arteriosclerosis. 1990 Sep-Oct;10(5):727-31. doi: 10.1161/01.atv.10.5.727. PMID 2403300
- [Background] Haffner SM, Stern MP, Hazuda HP, Mitchell BD, Patterson JK. Cardiovascular risk factors in confirmed prediabetic individuals. Does the clock for coronary heart disease start ticking before the onset of clinical diabetes? JAMA. 1990 Jun 6;263(21):2893-8. doi: 10.1001/jama.263.21.2893. PMID 2338751
- [Background] Mitchell BD, Stern MP, Haffner SM, Hazuda HP, Patterson JK. Functional impairment in Mexican Americans and non-Hispanic whites with diabetes. J Clin Epidemiol. 1990;43(4):319-27. doi: 10.1016/0895-4356(90)90118-9. PMID 2324773
- [Background] Mitchell BD, Stern MP, Haffner SM, Hazuda HP, Patterson JK. Risk factors for cardiovascular mortality in Mexican Americans and non-Hispanic whites. San Antonio Heart Study. Am J Epidemiol. 1990 Mar;131(3):423-33. doi: 10.1093/oxfordjournals.aje.a115517. PMID 2301352
- [Background] Mitchell BD, Haffner SM, Hazuda HP, Patterson JK, Stern MP. Diabetes and coronary heart disease risk in Mexican Americans. Ann Epidemiol. 1992 Jan-Mar;2(1-2):101-6. doi: 10.1016/1047-2797(92)90043-p. PMID 1342250
- [Background] Gonzalez-Villalpando C, Stern MP, Villalpando E, Hazuda H, Haffner SM, Lisci E. [Prevalence of diabetes and glucose intolerance in a urban population at a low economic level]. Rev Invest Clin. 1992 Jul-Sep;44(3):321-8. Spanish. PMID 1488576
- [Background] Edelstein SL, Knowler WC, Bain RP, Andres R, Barrett-Connor EL, Dowse GK, Haffner SM, Pettitt DJ, Sorkin JD, Muller DC, Collins VR, Hamman RF. Predictors of progression from impaired glucose tolerance to NIDDM: an analysis of six prospective studies. Diabetes. 1997 Apr;46(4):701-10. doi: 10.2337/diab.46.4.701. PMID 9075814
- [Background] Mykkanen L, Haffner SM, Rainwater DL, Karhapaa P, Miettinen H, Laakso M. Relationship of LDL size to insulin sensitivity in normoglycemic men. Arterioscler Thromb Vasc Biol. 1997 Jul;17(7):1447-53. doi: 10.1161/01.atv.17.7.1447. PMID 9261279
- [Background] Haffner SM, Hanefeld M, Fischer S, Fucker K, Leonhardt W. Glibenclamide, but not acarbose, increases leptin concentrations parallel to changes in insulin in subjects with NIDDM. Diabetes Care. 1997 Sep;20(9):1430-4. doi: 10.2337/diacare.20.9.1430. PMID 9283792
- [Background] Gonzalez Villalpando C, Rivera Martinez D, Arredondo Perez B, Martinez Diaz S, Gonzalez Villalpando ME, Haffner SM, Stern MP. High prevalence of cholelithiasis in a low income Mexican population: an ultrasonographic survey. Arch Med Res. 1997 Winter;28(4):543-7. PMID 9428581
- [Background] Haffner SM, Miettinen H, Stern MP. The homeostasis model in the San Antonio Heart Study. Diabetes Care. 1997 Jul;20(7):1087-92. doi: 10.2337/diacare.20.7.1087. PMID 9203442
- [Background] Haffner SM, Mykkanen L, Stern MP. Leptin concentrations in women in the San Antonio Heart Study: effect of menopausal status and postmenopausal hormone replacement therapy. Am J Epidemiol. 1997 Oct 1;146(7):581-5. doi: 10.1093/oxfordjournals.aje.a009317. PMID 9326436
- [Background] Haffner SM, Miettinen H, Stern MP. Relatively more atherogenic coronary heart disease risk factors in prediabetic women than in prediabetic men. Diabetologia. 1997 Jun;40(6):711-7. doi: 10.1007/s001250050738. PMID 9222652
- [Background] Gonzalez Villalpando ME, Gonzalez Villalpando C, Arredondo Perez B, Martinez Diaz SV, Mitchell B, Rivera Martinez D, Klein R, Haffner SM, Stern MP. Moderate-to-severe diabetic retinopathy is more prevalent in Mexico City than in San Antonio, Texas. Diabetes Care. 1997 May;20(5):773-7. doi: 10.2337/diacare.20.5.773. PMID 9135941
- [Background] Haffner SM, Miettinen H, Stern MP. Are risk factors for conversion to NIDDM similar in high and low risk populations? Diabetologia. 1997 Jan;40(1):62-6. doi: 10.1007/s001250050643. PMID 9028719
- [Background] Wei M, Stern MP, Haffner SM. Serum leptin levels in Mexican Americans and non-Hispanic whites: association with body mass index and cigarette smoking. Ann Epidemiol. 1997 Feb;7(2):81-6. doi: 10.1016/s1047-2797(96)00114-7. PMID 9099395
- [Background] Wei M, Gaskill SP, Haffner SM, Stern MP. Waist circumference as the best predictor of noninsulin dependent diabetes mellitus (NIDDM) compared to body mass index, waist/hip ratio and other anthropometric measurements in Mexican Americans--a 7-year prospective study. Obes Res. 1997 Jan;5(1):16-23. doi: 10.1002/j.1550-8528.1997.tb00278.x. PMID 9061711
- [Background] Haffner SM, Miettinen H, Gaskill SP, Stern MP. Decreased insulin action and insulin secretion predict the development of impaired glucose tolerance. Diabetologia. 1996 Oct;39(10):1201-7. doi: 10.1007/BF02658507. PMID 8897008
- [Background] Haffner SM, Kennedy E, Gonzalez C, Stern MP, Miettinen H. A prospective analysis of the HOMA model. The Mexico City Diabetes Study. Diabetes Care. 1996 Oct;19(10):1138-41. doi: 10.2337/diacare.19.10.1138. PMID 8886564
- [Background] Pugh JA, Tuley MR, Hazuda HP, Stern MP. The influence of outpatient insurance coverage on the microvascular complications of non-insulin-dependent diabetes in Mexican Americans. J Diabetes Complications. 1992 Oct-Dec;6(4):236-41. doi: 10.1016/1056-8727(92)90058-s. PMID 1482781
- [Background] Haffner SM, Gruber KK, Morales PA, Hazuda HP, Valdez RA, Mitchell BD, Stern MP. Lipoprotein(a) concentrations in Mexican Americans and non-Hispanic whites: the San Antonio Heart Study. Am J Epidemiol. 1992 Nov 1;136(9):1060-8. doi: 10.1093/oxfordjournals.aje.a116571. PMID 1462966
- [Background] Stern MP, Morales PA, Haffner SM, Valdez RA. Hyperdynamic circulation and the insulin resistance syndrome ("syndrome X"). Hypertension. 1992 Dec;20(6):802-8. doi: 10.1161/01.hyp.20.6.802. PMID 1452296
- [Background] Haffner SM, Valdez R, Morales PA, Mitchell BD, Hazuda HP, Stern MP. Greater effect of glycemia on incidence of hypertension in women than in men. Diabetes Care. 1992 Oct;15(10):1277-84. doi: 10.2337/diacare.15.10.1277. PMID 1425089
- [Background] Haffner SM, Morales PA, Stern MP, Gruber MK. Lp(a) concentrations in NIDDM. Diabetes. 1992 Oct;41(10):1267-72. doi: 10.2337/diab.41.10.1267. PMID 1397699
- [Background] Stern MP, Mitchell BD, Haffner SM, Hazuda HP. Does glycemic control of type II diabetes suffice to control diabetic dyslipidemia? A community perspective. Diabetes Care. 1992 May;15(5):638-44. doi: 10.2337/diacare.15.5.638. PMID 1516483
- [Background] Haffner SM, Ferrannini E, Hazuda HP, Stern MP. Clustering of cardiovascular risk factors in confirmed prehypertensive individuals. Hypertension. 1992 Jul;20(1):38-45. doi: 10.1161/01.hyp.20.1.38. PMID 1618551
- [Background] Haffner SM, Valdez RA, Hazuda HP, Mitchell BD, Morales PA, Stern MP. Prospective analysis of the insulin-resistance syndrome (syndrome X). Diabetes. 1992 Jun;41(6):715-22. doi: 10.2337/diab.41.6.715. PMID 1587398
- [Background] Haffner SM, Stern MP, Watanabe RM, Bergman RN. Relationship of insulin clearance and secretion to insulin sensitivity in non-diabetic Mexican Americans. Eur J Clin Invest. 1992 Mar;22(3):147-53. doi: 10.1111/j.1365-2362.1992.tb01819.x. PMID 1582438
- [Background] Haffner SM, Mitchell BD, Valdez RA, Hazuda HP, Morales PA, Stern MP. Eight-year incidence of hypertension in Mexican-Americans and non-Hispanic whites. The San Antonio Heart Study. Am J Hypertens. 1992 Mar;5(3):147-53. doi: 10.1093/ajh/5.3.147. PMID 1575941
- [Background] Mitchell BD, Hazuda HP, Haffner SM, Patterson JK, Stern MP. High prevalence of angina pectoris in Mexican-American men. A population with reduced risk of myocardial infarction. Ann Epidemiol. 1991 Aug;1(5):415-26. doi: 10.1016/1047-2797(91)90011-z. PMID 1669522
- [Background] Haffner SM, Hazuda HP, Mitchell BD, Patterson JK, Stern MP. Increased incidence of type II diabetes mellitus in Mexican Americans. Diabetes Care. 1991 Feb;14(2):102-8. doi: 10.2337/diacare.14.2.102. PMID 2060411
- [Background] Mayer MN, de Montalembert M, Audat F, Brusset MC, Houfani B, Merckx J, Barrier G, Gazengel C. Autologous blood donation for elective surgery in children weighing 8-25 kg. Vox Sang. 1996;70(4):224-8. doi: 10.1111/j.1423-0410.1996.tb01331.x. PMID 9123928
- [Background] Haffner SM, Mitchell BD, Hazuda HP, Stern MP. Greater influence of central distribution of adipose tissue on incidence of non-insulin-dependent diabetes in women than men. Am J Clin Nutr. 1991 May;53(5):1312-7. doi: 10.1093/ajcn/53.5.1312. PMID 2021139
- [Background] Mitchell BD, Hazuda HP, Haffner SM, Patterson JK, Stern MP. Myocardial infarction in Mexican-Americans and non-Hispanic whites. The San Antonio Heart Study. Circulation. 1991 Jan;83(1):45-51. doi: 10.1161/01.cir.83.1.45. PMID 1984897
- [Background] Berkus MD, Stern MP, Mitchell BD, Abashawl A, Langer O. Relationships between glucose levels and insulin secretion during a glucose challenge test. Am J Obstet Gynecol. 1990 Dec;163(6 Pt 1):1818-22. doi: 10.1016/0002-9378(90)90756-w. PMID 2256488
- [Background] Stern MP, Patterson JK, Mitchell BD, Haffner SM, Hazuda HP. Overweight and mortality in Mexican Americans. Int J Obes. 1990 Jul;14(7):623-9. PMID 2228397
- [Background] Stern MP, Haffner SM. Type II diabetes and its complications in Mexican Americans. Diabetes Metab Rev. 1990 Feb;6(1):29-45. doi: 10.1002/dmr.5610060102. PMID 2192854
- [Background] Haffner SM, Mitchell BD, Stern MP, Hazuda HP, Patterson JK. Decreased prevalence of hypertension in Mexican-Americans. Hypertension. 1990 Sep;16(3):225-32; discussion 233-4. doi: 10.1161/01.hyp.16.3.225. PMID 2394482
- [Background] Haffner SM, Klein R, Moss SE, Klein BE. Sex hormones and the incidence of severe retinopathy in male subjects with type I diabetes. Ophthalmology. 1993 Dec;100(12):1782-6. doi: 10.1016/s0161-6420(93)31398-9. PMID 8259274
- [Background] Haffner SM, Agil A, Mykkanen L, Stern MP, Jialal I. Plasma oxidizability in subjects with normal glucose tolerance, impaired glucose tolerance, and NIDDM. Diabetes Care. 1995 May;18(5):646-53. doi: 10.2337/diacare.18.5.646. PMID 8586002
- [Background] Haffner SM, Mykkanen L, Robbins D, Valdez R, Miettinen H, Howard BV, Stern MP, Bowsher R. A preponderance of small dense LDL is associated with specific insulin, proinsulin and the components of the insulin resistance syndrome in non-diabetic subjects. Diabetologia. 1995 Nov;38(11):1328-36. doi: 10.1007/BF00401766. PMID 8582543
- [Background] Valdez R, Gonzalez-Villalpando C, Mitchell BD, Haffner SM, Stern MP. Differential impact of obesity in related populations. Obes Res. 1995 Sep;3 Suppl 2:223s-232s. doi: 10.1002/j.1550-8528.1995.tb00468.x. PMID 8581781
- [Background] Gonzalez C, Stern MP, Mitchell B, Arredondo B, Martinez S, Seoane M. Myocardial infarction in a low income area of Mexico City. Prevalence and clinical characteristics. Arch Med Res. 1995 Autumn;26(3):233-8. PMID 8580673
- [Background] Gonzalez-Villalpando C, Stern MP, Rivera Martinez D, Arredondo Perez B, Martinez Diaz S, Haffner S. Carotid artery atherosclerosis in a Mexico City population with high carbohydrate intake. Arch Med Res. 1995 Winter;26(4):409-13. PMID 8555736
- [Background] Monterrosa AE, Haffner SM, Stern MP, Hazuda HP. Sex difference in lifestyle factors predictive of diabetes in Mexican-Americans. Diabetes Care. 1995 Apr;18(4):448-56. doi: 10.2337/diacare.18.4.448. PMID 7497852
- [Background] Haffner SM, Gonzalez C, Miettinen H, Howard BV, Stern MP. LDL size and subclass pattern in Mexico City residents and San Antonio Mexican Americans. Arterioscler Thromb Vasc Biol. 1995 Dec;15(12):2136-41. doi: 10.1161/01.atv.15.12.2136. PMID 7489234
- [Background] Haffner SM, Miettinen H, Gaskill SP, Stern MP. Decreased insulin secretion and increased insulin resistance are independently related to the 7-year risk of NIDDM in Mexican-Americans. Diabetes. 1995 Dec;44(12):1386-91. doi: 10.2337/diab.44.12.1386. PMID 7589843
- [Background] Haffner SM, Stern MP, Miettinen H, Gingerich R, Bowsher RR. Higher proinsulin and specific insulin are both associated with a parental history of diabetes in nondiabetic Mexican-American subjects. Diabetes. 1995 Oct;44(10):1156-60. doi: 10.2337/diab.44.10.1156. PMID 7556950
- [Background] Valdez R, Howard BV, Stern MP, Haffner SM. Apolipoprotein E polymorphism and insulin levels in a biethnic population. Diabetes Care. 1995 Jul;18(7):992-1000. doi: 10.2337/diacare.18.7.992. PMID 7555562
- [Background] Sowers M, Gonzalez Villalpando C, Stern MP, Fox C, Mitchell BD. Relationships between physical activity, insulin levels and lipids in non-diabetic low income residents of Mexico City: the Mexico City Diabetes Study. Arch Med Res. 1995 Summer;26(2):133-40. PMID 7620278
- [Background] Wei M, Valdez RA, Mitchell BD, Haffner SM, Stern MP, Hazuda HP. Migration status, socioeconomic status, and mortality rates in Mexican Americans and non-Hispanic whites: the San Antonio Heart Study. Ann Epidemiol. 1996 Jul;6(4):307-13. doi: 10.1016/s1047-2797(96)00026-9. PMID 8876841
- [Background] Haffner SM, Gingerich RL, Miettinen H, Stern MP. Leptin concentrations in relation to overall adiposity and regional body fat distribution in Mexican Americans. Int J Obes Relat Metab Disord. 1996 Oct;20(10):904-8. PMID 8910093
- [Background] Wei M, Mitchell BD, Haffner SM, Stern MP. Effects of cigarette smoking, diabetes, high cholesterol, and hypertension on all-cause mortality and cardiovascular disease mortality in Mexican Americans. The San Antonio Heart Study. Am J Epidemiol. 1996 Dec 1;144(11):1058-65. doi: 10.1093/oxfordjournals.aje.a008878. PMID 8942437
- [Background] Wei M, Gonzalez C, Haffner SM, O'Leary DH, Stern MP. Ultrasonographically assessed maximum carotid artery wall thickness in Mexico City residents and Mexican Americans living in San Antonio, Texas. Association with diabetes and cardiovascular risk factors. Arterioscler Thromb Vasc Biol. 1996 Nov;16(11):1388-92. doi: 10.1161/01.atv.16.11.1388. PMID 8911278
- [Background] Gonzalez ME, Gonzalez C, Stern MP, Arredondo B, Martinez S. Concordance in diagnosis of diabetic retinopathy by fundus photography between retina specialists and a standardized reading center. Mexico City Diabetes Study Retinopathy Group. Arch Med Res. 1995 Summer;26(2):127-31. PMID 7620277
- [Background] Mitchell BD, Gonzalez Villalpando C, Arredondo Perez B, Garcia MS, Valdez R, Stern MP. Myocardial infarction and cardiovascular risk factors in Mexico City and San Antonio, Texas. Arterioscler Thromb Vasc Biol. 1995 Jun;15(6):721-5. doi: 10.1161/01.atv.15.6.721. PMID 7773724
- [Background] Gonzalez Villalpando C, Stern MP, Arredondo Perez B, Martinez Diaz S. The level of metabolic control in low income Mexico City Diabetics. The Mexico City Diabetes Study. Arch Med Res. 1994 Winter;25(4):387-92. PMID 7858396
- [Background] Haffner SM, Mykkanen L, Stern MP, Paidi M, Howard BV. Greater effect of diabetes on LDL size in women than in men. Diabetes Care. 1994 Oct;17(10):1164-71. doi: 10.2337/diacare.17.10.1164. PMID 7821137
- [Background] Gonzalez Villalpando ME, Gonzalez Villalpando C, Arredondo Perez B, Stern MP. Diabetic retinopathy in Mexico. Prevalence and clinical characteristics. Arch Med Res. 1994 Autumn;25(3):355-60. PMID 7803988
- [Background] Gonzalez Villalpando C, Stern MP, Arredondo Perez B, Valdez R, Mitchell B, Haffner S. Prevalence and detection of hypertension in Mexico. Arch Med Res. 1994 Autumn;25(3):347-53. PMID 7803987
- [Background] Haffner SM, Mykkanen L, Valdez RA, Stern MP, Holloway DL, Monterrosa A, Bowsher RR. Disproportionately increased proinsulin levels are associated with the insulin resistance syndrome. J Clin Endocrinol Metab. 1994 Dec;79(6):1806-10. doi: 10.1210/jcem.79.6.7989488.
- [Background] Gonzalez-Villalpando C, Stern MP, Arredondo-Perez B. [The use of hospital services by diabetic patients: study in an open population]. Salud Publica Mex. 1994 Jul-Aug;36(4):415-9. Spanish. PMID 7973995
- [Background] Haffner SM, Bowsher RR, Mykkanen L, Hazuda HP, Mitchell BD, Valdez RA, Gingerich R, Monterossa A, Stern MP. Proinsulin and specific insulin concentration in high- and low-risk populations for NIDDM. Diabetes. 1994 Dec;43(12):1490-3. doi: 10.2337/diab.43.12.1490. PMID 7958504
- [Background] Valdez R, Athens MA, Thompson GH, Bradshaw BS, Stern MP. Birthweight and adult health outcomes in a biethnic population in the USA. Diabetologia. 1994 Jun;37(6):624-31. doi: 10.1007/BF00403383. PMID 7926349
- [Background] Haffner SM, Mykkanen L, Valdez RA, Stern MP. Evaluation of two insulin assays in insulin resistance syndrome (syndrome X). Arterioscler Thromb. 1994 Sep;14(9):1430-7. doi: 10.1161/01.atv.14.9.1430. PMID 8068604
- [Background] Gonzelez C, Stern MP, Mitchell BD, Valdez RA, Haffner SM, Perez BA. Clinical characteristics of type II diabetic subjects consuming high versus low carbohydrate diets in Mexico City and San Antonio, Texas. Diabetes Care. 1994 May;17(5):397-404. doi: 10.2337/diacare.17.5.397. PMID 8062606
- [Background] Haffner SM, Valdez RA, Mykkanen L, Stern MP, Katz MS. Decreased testosterone and dehydroepiandrosterone sulfate concentrations are associated with increased insulin and glucose concentrations in nondiabetic men. Metabolism. 1994 May;43(5):599-603. doi: 10.1016/0026-0495(94)90202-x. PMID 8177048
- [Background] Valdez R, Mitchell BD, Haffner SM, Hazuda HP, Morales PA, Monterrosa A, Stern MP. Predictors of weight change in a bi-ethnic population. The San Antonio Heart Study. Int J Obes Relat Metab Disord. 1994 Feb;18(2):85-91. PMID 8148929
- [Background] Haffner SM, Mitchell BD, Moss SE, Stern MP, Hazuda HP, Patterson J, Van Heuven WA, Klein R. Is there an ethnic difference in the effect of risk factors for diabetic retinopathy? Ann Epidemiol. 1993 Jan;3(1):2-8. doi: 10.1016/1047-2797(93)90003-m. PMID 8287152
- [Background] Haffner SM, Valdez RA, Stern MP, Katz MS. Obesity, body fat distribution and sex hormones in men. Int J Obes Relat Metab Disord. 1993 Nov;17(11):643-9. PMID 8281222
- [Background] Stern MP, Gonzalez C, Hernandex M, Knapp JA, Hazuda HP, Villapando E, Valdez RA, Haffner SM, Mitchell BD. Performance of semiquantitative food frequency questionnaires in international comparisons. Mexico City versus San Antonio, Texas. Ann Epidemiol. 1993 May;3(3):300-7. doi: 10.1016/1047-2797(93)90034-2. PMID 8275204
- [Background] Haffner SM, Gonzales C, Valdez RA, Mykkanen L, Hazuda HP, Mitchell BD, Monterrosa A, Stern MP. Is microalbuminuria part of the prediabetic state? The Mexico City Diabetes Study. Diabetologia. 1993 Oct;36(10):1002-6. doi: 10.1007/BF02374491. PMID 8243847
- [Background] Haffner SM, Mykkanen L, Valdez RA, Paidi M, Stern MP, Howard BV. LDL size and subclass pattern in a biethnic population. Arterioscler Thromb. 1993 Nov;13(11):1623-30. doi: 10.1161/01.atv.13.11.1623. PMID 8218103
- [Background] Haffner SM, Diehl AK, Valdez R, Mitchell BD, Hazuda HP, Morales P, Stern MP. Clinical gallbladder disease in NIDDM subjects. Relationship to duration of diabetes and severity of glycemia. Diabetes Care. 1993 Sep;16(9):1276-84. doi: 10.2337/diacare.16.9.1276. PMID 8404432
- [Background] Mitchell BD, Valdez R, Hazuda HP, Haffner SM, Monterrosa A, Stern MP. Differences in the prevalence of diabetes and impaired glucose tolerance according to maternal or paternal history of diabetes. Diabetes Care. 1993 Sep;16(9):1262-7. doi: 10.2337/diacare.16.9.1262. PMID 8404430
- [Background] Stern MP, Valdez RA, Haffner SM, Mitchell BD, Hazuda HP. Stability over time of modern diagnostic criteria for type II diabetes. Diabetes Care. 1993 Jul;16(7):978-83. doi: 10.2337/diacare.16.7.978. PMID 8359106
- [Background] Haffner SM, Mykkanen L, Stern MP, Valdez RA, Heisserman JA, Bowsher RR. Relationship of proinsulin and insulin to cardiovascular risk factors in nondiabetic subjects. Diabetes. 1993 Sep;42(9):1297-302. doi: 10.2337/diab.42.9.1297. PMID 8349041
- [Background] Gonzalez Villalpando C, Stern MP, Valdez R, Mitchell B, Haffner S. [Blood lipid levels and atherogenic risk in an open urban population]. Rev Invest Clin. 1993 Mar-Apr;45(2):127-32. Spanish. PMID 8337539
- [Background] Haffner SM, Valdez RA, Morales PA, Hazuda HP, Stern MP. Decreased sex hormone-binding globulin predicts noninsulin-dependent diabetes mellitus in women but not in men. J Clin Endocrinol Metab. 1993 Jul;77(1):56-60. doi: 10.1210/jcem.77.1.8325960.
- [Background] Kariakin AM, Aliev SA, Ivanov MA. [Our experience and the outlook for the development of surgery in esophageal cancer]. Vestn Khir Im I I Grek. 1997;156(3):64-7. Russian. PMID 9324849
- [Background] Stern MP, Morales PA, Valdez RA, Monterrosa A, Haffner SM, Mitchell BD, Hazuda HP. Predicting diabetes. Moving beyond impaired glucose tolerance. Diabetes. 1993 May;42(5):706-14. doi: 10.2337/diab.42.5.706. PMID 8482427
- [Background] Haffner SM, Morales PA, Gruber MK, Hazuda HP, Stern MP. Cardiovascular risk factors in non-insulin-dependent diabetic subjects with microalbuminuria. Arterioscler Thromb. 1993 Feb;13(2):205-10. doi: 10.1161/01.atv.13.2.205. PMID 8427856
- [Background] Morales PA, Mitchell BD, Valdez RA, Hazuda HP, Stern MP, Haffner SM. Incidence of NIDDM and impaired glucose tolerance in hypertensive subjects. The San Antonio Heart Study. Diabetes. 1993 Jan;42(1):154-61. doi: 10.2337/diab.42.1.154. PMID 8420812
- [Background] Haffner SM, Morales PA, Hazuda HP, Stern MP. Level of control of hypertension in Mexican Americans and non-Hispanic whites. Hypertension. 1993 Jan;21(1):83-8. doi: 10.1161/01.hyp.21.1.83. PMID 8418027
- [Background] Gonzalez Villalpando C, Stern MP, Arredondo Perez B, Martinez Diaz S, Islas Andrade S, Revilla C, Gonzalez Villalpando ME, Rivera Martinez D. Nephropathy in low income diabetics: the Mexico City Diabetes Study. Arch Med Res. 1996 Autumn;27(3):367-72. PMID 8854397
- [Background] Haffner SM, Miettinen H, Gaskill SP, Stern MP. Metabolic precursors of hypertension. The San Antonio Heart Study. Arch Intern Med. 1996 Sep 23;156(17):1994-2001. PMID 8823152
- [Background] Gonzalez Villalpando C, Stern MP, Arredondo Perez B, Martinez Diaz S, Haffner S. Undiagnosed hypercholesterolemia: a serious health challenge. The Mexico City Diabetes Study. Arch Med Res. 1996 Spring;27(1):19-23. PMID 8867362
- [Background] Haffner SM, Stern MP, Miettinen H, Robbins D, Howard BV. Apolipoprotein E polymorphism and LDL size in a biethnic population. Arterioscler Thromb Vasc Biol. 1996 Sep;16(9):1184-8. doi: 10.1161/01.atv.16.9.1184. PMID 8792773
- [Background] Gonzalez Villalpando C, Stern MP, Arredondo Perez B, Martijnez Diaz S, Gonzalez Villalpando ME, Haffner S, Rivera D, Diehl AK. Prevalence of gallbladder disease and associated clinical variables in a low income population of Mexico City. Arch Med Res. 1996 Summer;27(2):237-41. PMID 8696071
- [Background] Gonzalez ME, Gonzalez C, Stern MP, Arredondo B, Martinez Diaz S. Concordance between retina specialists and a preferred practice pattern in treatment and follow-up criteria for diabetic retinopathy. The Mexico City Diabetes Study Retinopathy Group. Arch Med Res. 1996 Summer;27(2):205-11. PMID 8696066
- [Background] Haffner SM, Miettinen H, Stern MP, Agil A, Jialal I. Plasma oxidizability in Mexican-Americans and non-Hispanic whites. Metabolism. 1996 Jul;45(7):876-81. doi: 10.1016/s0026-0495(96)90163-8. PMID 8692025
- [Background] Duggirala R, Gonzalez Villalpando C, O'Leary DH, Stern MP, Blangero J. Genetic basis of variation in carotid artery wall thickness. Stroke. 1996 May;27(5):833-7. doi: 10.1161/01.str.27.5.833. PMID 8623101
- [Background] Stern MP, Wei M. Do Mexican Americans really have low rates of cardiovascular disease? Prev Med. 1999 Dec;29(6 Pt 2):S90-5. doi: 10.1006/pmed.1998.0464. PMID 10641824
- [Background] Gonzalez-Villalpando C, Gonzalez-Villalpando ME, Rivera Martinez D, Stern MP. [Incidence and progression of diabetic retinopathy in low income population of Mexico City]. Rev Invest Clin. 1999 May-Jun;51(3):141-50. Spanish. PMID 10466004
- [Background] Gonzalez-Villalpando C, Stern MP, Haffner SM, Gonzalez Villapando ME, Gaskill S, Rivera Martinez D. Prevalence of hypertension in a Mexican population according to the Sixth Report of the Joint National Committee on Prevention, Detection, Evaluation and Treatment of High Blood Pressure. J Cardiovasc Risk. 1999 Jun;6(3):177-81. doi: 10.1177/204748739900600309. PMID 10463145
- [Background] Gonzalez C, Stern MP, Gonzalez E, Rivera D, Simon J, Islas S, Haffner S. The Mexico City Diabetes Study: a population-based approach to the study of genetic and environmental interactions in the pathogenesis of obesity and diabetes. Nutr Rev. 1999 May;57(5 Pt 2):S71-6; discussion S76-7. doi: 10.1111/j.1753-4887.1999.tb01792.x. No abstract available. PMID 10391030
- [Background] Haffner SM, Miettinen H, Mykkanen L, Stern MP. Leptin concentrations are associated with higher proinsulin and insulin concentrations but a lower proinsulin/insulin ratio in non-diabetic subjects. Int J Obes Relat Metab Disord. 1998 Sep;22(9):899-905. doi: 10.1038/sj.ijo.0800679. PMID 9756249
- [Background] Haffner SM, Mykkanen LA, Gonzalez CC, Stern MP. Leptin concentrations do not predict weight gain: the Mexico City Diabetes Study. Int J Obes Relat Metab Disord. 1998 Jul;22(7):695-9. doi: 10.1038/sj.ijo.0800619. PMID 9705032
- [Background] Wei M, Gibbons LW, Mitchell TL, Kampert JB, Stern MP, Blair SN. Low fasting plasma glucose level as a predictor of cardiovascular disease and all-cause mortality. Circulation. 2000 May 2;101(17):2047-52. doi: 10.1161/01.cir.101.17.2047. PMID 10790345
- [Background] Burke JP, Williams K, Gaskill SP, Hazuda HP, Haffner SM, Stern MP. Rapid rise in the incidence of type 2 diabetes from 1987 to 1996: results from the San Antonio Heart Study. Arch Intern Med. 1999 Jul 12;159(13):1450-6. doi: 10.1001/archinte.159.13.1450. PMID 10399896
- [Background] Lorenzo C, Serrano-Rios M, Martinez-Larrad MT, Gabriel R, Williams K, Gonzalez-Villalpando C, Stern MP, Hazuda HP, Haffner S. Prevalence of hypertension in Hispanic and non-Hispanic white populations. Hypertension. 2002 Feb;39(2):203-8. doi: 10.1161/hy0202.103439. PMID 11847184
- [Background] Lorenzo C, Serrano-Rios M, Martinez-Larrad MT, Gabriel R, Williams K, Gonzalez-Villalpando C, Stern MP, Hazuda HP, Haffner SM. Was the historic contribution of Spain to the Mexican gene pool partially responsible for the higher prevalence of type 2 diabetes in mexican-origin populations? The Spanish Insulin Resistance Study Group, the San Antonio Heart Study, and the Mexico City Diabetes Study. Diabetes Care. 2001 Dec;24(12):2059-64. doi: 10.2337/diacare.24.12.2059. PMID 11723083
- [Background] Burke JP, Williams K, Haffner SM, Villalpando CG, Stern MP. Elevated incidence of type 2 diabetes in San Antonio, Texas, compared with that of Mexico City, Mexico. Diabetes Care. 2001 Sep;24(9):1573-8. doi: 10.2337/diacare.24.9.1573. PMID 11522701
- [Background] Stern MP, Williams K, Haffner SM. Identification of persons at high risk for type 2 diabetes mellitus: do we need the oral glucose tolerance test? Ann Intern Med. 2002 Apr 16;136(8):575-81. doi: 10.7326/0003-4819-136-8-200204160-00006. PMID 11955025
- [Background] Han TS, Sattar N, Williams K, Gonzalez-Villalpando C, Lean ME, Haffner SM. Prospective study of C-reactive protein in relation to the development of diabetes and metabolic syndrome in the Mexico City Diabetes Study. Diabetes Care. 2002 Nov;25(11):2016-21. doi: 10.2337/diacare.25.11.2016. PMID 12401749
- [Background] Stern MP, Fatehi P, Williams K, Haffner SM. Predicting future cardiovascular disease: do we need the oral glucose tolerance test? Diabetes Care. 2002 Oct;25(10):1851-6. doi: 10.2337/diacare.25.10.1851. PMID 12351490
- [Background] Hanley AJ, Williams K, Gonzalez C, D'Agostino RB Jr, Wagenknecht LE, Stern MP, Haffner SM; San Antonio Heart Study; Mexico City Diabetes Study; Insulin Resistance Atherosclerosis Study. Prediction of type 2 diabetes using simple measures of insulin resistance: combined results from the San Antonio Heart Study, the Mexico City Diabetes Study, and the Insulin Resistance Atherosclerosis Study. Diabetes. 2003 Feb;52(2):463-9. doi: 10.2337/diabetes.52.2.463. PMID 12540622
- [Background] Del Rincon I, Williams K, Stern MP, Freeman GL, O'Leary DH, Escalante A. Association between carotid atherosclerosis and markers of inflammation in rheumatoid arthritis patients and healthy subjects. Arthritis Rheum. 2003 Jul;48(7):1833-40. doi: 10.1002/art.11078. PMID 12847676
- [Background] Burke JP, Williams K, Narayan KM, Leibson C, Haffner SM, Stern MP. A population perspective on diabetes prevention: whom should we target for preventing weight gain? Diabetes Care. 2003 Jul;26(7):1999-2004. doi: 10.2337/diacare.26.7.1999. PMID 12832302
- [Background] Hunt KJ, Williams K, Resendez RG, Hazuda HP, Haffner SM, Stern MP. All-cause and cardiovascular mortality among diabetic participants in the San Antonio Heart Study: evidence against the "Hispanic Paradox". Diabetes Care. 2002 Sep;25(9):1557-63. doi: 10.2337/diacare.25.9.1557. PMID 12196427
- [Background] Hunt KJ, Resendez RG, Williams K, Haffner SM, Stern MP, Hazuda HP. All-cause and cardiovascular mortality among Mexican-American and non-Hispanic White older participants in the San Antonio Heart Study- evidence against the "Hispanic paradox". Am J Epidemiol. 2003 Dec 1;158(11):1048-57. doi: 10.1093/aje/kwg249. PMID 14630600
- [Background] Hunt KJ, Williams K, Rivera D, O'Leary DH, Haffner SM, Stern MP, Gonzalez Villalpando C. Elevated carotid artery intima-media thickness levels in individuals who subsequently develop type 2 diabetes. Arterioscler Thromb Vasc Biol. 2003 Oct 1;23(10):1845-50. doi: 10.1161/01.ATV.0000093471.58663.ED. Epub 2003 Sep 4. PMID 12958039
- [Background] Meigs JB, Williams K, Sullivan LM, Hunt KJ, Haffner SM, Stern MP, Gonzalez Villalpando C, Perhanidis JS, Nathan DM, D'Agostino RB Jr, D'Agostino RB Sr, Wilson PW. Using metabolic syndrome traits for efficient detection of impaired glucose tolerance. Diabetes Care. 2004 Jun;27(6):1417-26. doi: 10.2337/diacare.27.6.1417. PMID 15161798
- [Background] Hunt KJ, Resendez RG, Williams K, Haffner SM, Stern MP; San Antonio Heart Study. National Cholesterol Education Program versus World Health Organization metabolic syndrome in relation to all-cause and cardiovascular mortality in the San Antonio Heart Study. Circulation. 2004 Sep 7;110(10):1251-7. doi: 10.1161/01.CIR.0000140762.04598.F9. Epub 2004 Aug 23. PMID 15326061
- [Background] Mitchell BD, Haffner SM, Hazuda HP, Valdez R, Stern MP. The relation between serum insulin levels and 8-year changes in lipid, lipoprotein, and blood pressure levels. Am J Epidemiol. 1992 Jul 1;136(1):12-22. doi: 10.1093/oxfordjournals.aje.a116416. PMID 1415128
- [Background] Stern MP, Gonzalez C, Mitchell BD, Villalpando E, Haffner SM, Hazuda HP. Genetic and environmental determinants of type II diabetes in Mexico City and San Antonio. Diabetes. 1992 Apr;41(4):484-92. doi: 10.2337/diab.41.4.484. PMID 1607073
- [Background] Gonzalez-Villalpando C, Stern MP, Arredondo-Perez B, Mitchell B, Valdez R, Haffner S. [Tobacco use in Mexico City]. Salud Publica Mex. 1994 Jan-Feb;36(1):46-50. Spanish. PMID 8042071